CLINICAL TRIAL: NCT06767865
Title: Online Diabetes Clinic Support Program for Type 2 Diabetic Individuals New to Insulin Therapy
Brief Title: Online Diabetes Clinic Support Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilek Büyükkaya Besen (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Dilek Büyükkaya Besen, Assoc. Prof., Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DokuzEU-IHH-DBB-01
Record Dates: First submitted 2024-12-30; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Endocrine System Diseases; Education; Nursing Education
Keywords: Insulin therapy; online clinic; continuous support and follow-up; type 2 diabetes
MeSH Terms: conditions — Endocrine System Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Individuals in the experimental group received online training and were subsequently provided with continuous follow-up, counseling, motivation and informative message support for three months. In addition, patients were given a target board containing a daily diabetes management program and were asked to use it for three months.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): intervention+ Follow-up at 0-3-6 months
  Interventions: Other: online support programe
- Control Group (No Intervention): Follow-up at 0-3-6 months

INTERVENTIONS:
Other: online support programe — Individuals in the experimental group received online training and were subsequently provided with continuous follow-up, counseling, motivation and informative message support for three months. In addition, patients were given a target board containing a daily diabetes management program and were asked to use it for three months.
  Arms: Experimental Group

SUMMARY:
This study highlights the potential of online diabetes clinic support programs in improving treatment adherence, reducing treatment-related anxiety, and enhancing self-management skills in insulin therapy. Telehealth interventions play a crucial role in optimizing diabetes care and supporting patients in managing their insulin treatment effectively.

DETAILED DESCRIPTION:
This study was conducted to examine the effects of the online diabetes polyclinic continuous support program applied to individuals with type 2 diabetes who had just started insulin treatment on patient outcomes (metabolic, psychological and social parameters). The study was designed as a randomized controlled trial. It was conducted with 35 individuals in the experimental group who had just started insulin treatment and 32 individuals in the control group. Individuals were assessed with the individual diagnosis form, hypoglycemic confidence scale, hypoglycemia fear scale, diabetes empowerment scale short form, psychological insulin resistance scale, insulin treatment evaluation scale, perceived social support scale and diabetes history (treatment changes, HbA1c, lipid levels, frequency of hypoglycemia and hyperglycemia, frequency of emergency and hospital visits) before the intervention and in the 3rd and 6th months after the intervention. Individuals in the experimental group received online training and were subsequently provided with continuous follow-up, counseling, motivation and information-providing message support for three months. In addition, patients were given a target board containing a daily diabetes management program and were asked to use it for three months. As a result, it was determined that the online polyclinic service reduced the frequency of hypoglycemia and hyperglycemia in individuals who had just started insulin treatment and reduced emergency room visits (p<0.001). It was determined that it caused a significant decrease in the HbA1c and lipid levels of the patients in the experimental group and contributed to the cessation of insulin treatment under the supervision of a physician. It was determined that the online diabetes polyclinic continuous support program was effective in reducing hypoglycemia fear and psychological insulin resistance, and increased hypoglycemic confidence and empowerment levels (p<0.001). The study showed the potential of the online diabetes polyclinic continuous support initiative in improving the treatment process in patients who had just started insulin. These results reveal that online support systems can be effective in increasing patients' compliance with treatment and in better managing the treatment process. Online support has been shown to improve adherence to insulin therapy by providing patients with faster access to information, reduced anxiety about treatment, and greater self-management skills. This suggests that telehealth and online support programs may play an important role in diabetes management and insulin therapy acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and over,
* able to communicate in Turkish,
* diagnosed with type 2 diabetes,
* newly started insulin treatment,
* having and using information technology products (telephone, computer)
* willing to participate in the study voluntarily were included in the study.

Exclusion Criteria:

* Individuals with visual,
* auditory or cognitive impairments,
* a condition that prevents communication,
* cannot use information technology products,
* individuals who do not meet the inclusion criteria
* those who do not agree to participate in the study were not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Hypoglycemic Confidence Scale | 1 month
  The Hypoglycemic Confidence Scale is a nine-item self-report scale developed by William Polonsky and colleagues in 2017 that examines the degree to which diabetic patients feel confident and comfortable about their ability to avoid hypoglycemia-related problems. It was developed for use in adults with diabetes (Type 1 and Type 2 who use insulin). The Hypoglycemic Confidence Scale focuses on three areas: 1. Self-confidence (e.g., confidence in recognizing and managing hypoglycemia before blood sugar drops too low) 2. Confidence in avoiding hypoglycemia at critical times (e.g., while driving, exercising, and sleeping) 3. Estimation of spouse/partner's confidence. The Hypoglycemic Confidence Scale items are scored between 1-4 (1; Not at all confident 2; Somewhat confident 3; Moderately confident 4; Very confident). The ninth scale item for diabetic individuals with a spouse is interpreted as: 1; Not at all confident 2; Somewhat confident 3; Moderately confident 4; Very confident.
Hypoglycemia Fear Survey (HFS): | 1 month
  The Hypoglycemia Fear Survey- HFS, was used to determine the fear of hypoglycemia in diabetic individuals. This scale consists of two subgroups, behavior and anxiety, and a total of 33 items. The behavior subgroup of this scale consists of 15 items. In the behavior subgroup; diabetic individuals are asked about what they have done in their daily lives to prevent their blood glucose levels from falling in the last 6 months. The anxiety subgroup consists of 18 items, and individuals are asked how often they have worried about the items given due to the decrease in their blood glucose levels in the last 6 months. The answers range from; "0 points: never; 1 point: rarely; 2 points: sometimes; 3 points often; 4 points: always". The high score obtained indicates that the fear of hypoglycemia is high. The Turkish validity and reliability were made by Özgül Erol.
Diabetes Empowerment Scale (DES-Short Form): | 1 month
  The validity and reliability of the scale were made in 2020. DES-SF was designed to assess the empowerment levels of individuals regarding their health status. The scale is a five-point Likert type and has eight items (scored between "Strongly disagree" = 1 and "Strongly agree = 5"). The scale does not have a cut-off score. The scale is calculated based on the average score. An increase in the average score indicates an increase in the empowerment level.
Psychological Insulin Resistance Scale (PIRS) | 1 month
  The scale was developed by Song and colleagues in 2016. The scale, which is a 5-point Likert type (1: strongly agree, 2: agree, 3: undecided, 4: disagree, 5: strongly disagree), consists of 18 items and 2 sub-dimensions (Supportive factor and Psycho-cognitive/physical factor). The total score of the scale varies between 18-90. A high score obtained from the scale indicates that the patient's psychological resistance to insulin use is high. The scale was developed by Işık and Colleagues in 2021. As a result of the Turkish validity and reliability analysis, the scale consists of 12 items and 3 sub-dimensions (supportive, psycho-cognitive, physical factors). Cronbach's alpha coefficient was determined as 0.82.
Insulin Therapy Assessment Scale (ITAS) | 1 month
  The scale was developed by Sürücü et al. in 2017. Number of sub-dimensions and items: It consists of two sub-dimensions and a total of 20 items. Positive attitude (4 items): Items 3, 8, 17 and 19; Negative attitude (16 items): Items 1, 2, 4, 5, 6, 7, 9, 10, 11, 12, 13, 14, 15, 16, 18 and 20. Scale items are rated on a Likert type scale between "strongly disagree" and "strongly agree" and 5 points. The sum of four positively worded items (4-20) gives the positive evaluation sub-dimension, and the sum of 16 negatively worded items (16-80) gives the negative evaluation sub-dimension. The sum of the items (20 items) gives the total score (20-100). The scale total score is found by reversing the four positively worded items and summing them with the other 16 negatively worded items.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek D Büyükkaya Besen, PhD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, Izmir, Alsancak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No